CLINICAL TRIAL: NCT03486886
Title: PSMA-PET Imaging in Patients With Metastatic Prostate Cancer: Institutional Evaluation of Detection Yield Performance and Reproducibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17.068
Record Dates: First submitted 2018-03-19; First posted 2018-04-03 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA -PET/CT scanning (Experimental)
  Interventions: Diagnostic Test: PSMA -PET/CT scanning

INTERVENTIONS:
Diagnostic Test: PSMA -PET/CT scanning — PET/CT scanning is performed on hybrid PET/CT scanners. Patients should fast for at least 4 hours to facilitate transit of oral contrast into the distal small bowel. An oral contrast product can be administered and [18F]-DCFPyL is injected by IV rapid bolus followed by saline flush. 80-100 minutes following [18F]-DCFPyL injection, CT and PET images are consecutively acquired from the base of the skull to the upper thighs. An MRI of the questioned lesion sites may be performed.
  Uptake of lesions is measured with SUVmax. Hepatic and blood pool SUV is determined for the computation of tumor-to-liver and tumor-to-blood ratios.
  15 patients max will undergo a second PSMA-PET scan on the same camera with the same protocol using a different tracer batch within 2 weeks of the initial PSMA-PET evaluation in order to determine test-retest repeatability of the imaging procedure using a Bland-Altman analysis (per lesion analysis).

SUMMARY:
A promising imaging technique involving new prostate specific membrane antigen (PSMA) positron emission tomography (PET) tracers is emerging in metastatic prostate cancer (PCa). This approach has demonstrated higher sensitivity in detecting metastases, prior to and during therapy, than current imaging standard of care (CT and bone scan).

PSMA is expressed in the vast majority of PCa tissue specimens and its degree of expression correlates with a number of important metrics of PCa tumor aggressiveness.

[18F]DCFPyL is a promising high-sensitivity second generation PSMA-targeted urea-based PET probe. Studies employing second-generation PSMA PET/CT imaging in men with biochemical progression after definitive therapy suggest detection of metastases in over 60% of men imaged. In fact, PSMA-based PET has so far proven to have higher sensitivity than any other modality for localization of the site of recurrence. Applications that show promise and require further investigation include the characterization and risk stratification of primary PCa, complete staging of metastatic PCa to allow for PSMA-targeted radiotherapy and improved identification of patients with oligometastatic disease.

The objective of this study is to explore the detection yield of PSMA-PET in a pilot cohort of patients at CHUM and establish the repeatability of the technique before investigating it more widely.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Metastatic prostate cancer.
* At least 18 years of age
* Standard imaging (bone scan, CT abdo/pelvis/chest) within 6 weeks of consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Metastasis detection yield | 6 weeks
  Evaluation of the metastasis detection yield between PSMA PET/CT and standard imaging.

SECONDARY OUTCOMES:
Reproducibility of PSMA radiotracer uptake | 2 weeks
  Measure the repeatability of PSMA PET/CT imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada